CLINICAL TRIAL: NCT03130439
Title: A Phase 2 Study of Abemaciclib for Patients With Retinoblastoma-Positive, Triple Negative Metastatic Breast Cancer
Brief Title: Abemaciclib for Patients With Retinoblastoma-Positive, Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-024
Record Dates: First submitted 2017-04-24; First posted 2017-04-26 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib (Experimental): -Abemaciclib will be administered orally, twice daily on days 1 to 28
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib (LY2835219) has been shown in vitro to be a selective ATP-competitive inhibitor of CDK4 and CDK6 kinase activity that prevents the phosphorylation and subsequent inactivation of the Rb tumor suppressor protein, thereby inducing G1 cell cycle arrest and inhibition of cell proliferation.
  Other Names: LY2835219

SUMMARY:
This research study is studying a drug called Abemaciclib as a possible treatment for have metastatic triple-negative type of breast cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved abemaciclib as a treatment for any disease.

Some triple-negative breast cancers show expression of the Rb protein and are referred to as "Rb-positive." The Rb protein is important because it controls the way that cancer cells divide and grow. Drugs like abemaciclib work by changing the way that Rb functions. This can potentially stop cancer cells from dividing, and can also potentially lead to cancer cell death.

In this research study, the investigators are are looking to see how safe abemaciclib is and how well it will work to help people with triple-negative breast cancer that is Rb-positive.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, which is recurrent, locally advanced, unresectable or metastatic.
* Patients must have at least one lesion that is not within a previously radiated field and that is measurable on computerized tomography (CT) or magnetic resonance imaging (MRI) scans per RECIST version 1.1. Bone lesions are not considered measurable.
* Either the primary tumor and/or metastatic tumor must be triple-negative on the most recent sample as defined below:

  * Hormone receptor status: the invasive tumor must be ER- and PR-negative, or staining present in <1% by immunohistochemistry (IHC)
  * HER2 status: the invasive tumor must be Human Epidermal Growth Factor Receptor 2 Negative (HER2-negative) by the ASCO CAP guidelines
* Either the primary tumor and/or the metastatic tumor must be RB positive as defined below:

  --RB status: the invasive tumor must have greater than 50% of tumor cells staining positive for RB.
* Prior Chemotherapy:

  * Patients may have received 1-3 prior systemic therapies for metastatic disease (note: for patients who have first developed recurrent/metastatic disease within 12 months of completing any (neo)-adjuvant therapy for triple-negative breast cancer, the (neo)-adjuvant therapy is counted as a prior line of therapy).
  * Patients must have been off treatment with myelosuppressive chemotherapy for at least 21 days or nonmyelosuppressive agents for 14 days before registration. Patients should also be adequately recovered (to baseline or grade 1) from acute toxicities of prior treatment except for residual alopecia and peripheral neuropathy.
* Prior biologic therapy: Patients must have discontinued all biologic therapy at least 21 days before registration.
* Prior radiation therapy: Patients may have received prior radiation therapy in either the metastatic or early-stage setting. Radiation therapy must be completed at least 14 days prior to study registration.
* Patients on bisphosphonates or RANK-L inhibitors may continue receiving these therapies during study treatment. There is no washout period required between the last dose of these therapies and the start of abemaciclib.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1500/mm3
  * Platelets ≥100,000/mm3
  * Hemoglobin ≥8 g/dL
  * Total Bilirubin ≤1.5x the upper limit of normal (ULN)
  * Serum creatinine ≤1.5 mg/dL OR calculated GFR ≥60mL/min
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times the upper limit of normal. For patients with documented liver metastases, AST/ALT ≤ 5.0 times the upper limit of normal.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening. Women of childbearing potential are defined as those who have not been surgically sterilized and have had a menstrual period in the past year
* The patient must be ≥18 years old
* Capable of understanding and complying with the protocol and has signed the informed consent document.
* Able to swallow study drug.
* Sexually active patients (male and female) must use medically acceptable methods of contraception during the course of the study and for 3 months after completion of study treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately. While on the study and for 3 months after final drug administration, women may not breast-feed.
* Confirmed availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue
* Patients with tumor that is felt to be accessible to biopsy must be willing to provide tissue from a newly obtained core biopsy of a tumor lesion at baseline. Biopsies will be obtained up to 1 week (7 days) prior to initiation of treatment on Cycle 1, Day 1. Patients who undergo an attempted research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are not required to undergo a repeat biopsy in order to continue on protocol.

Exclusion Criteria:

* Received a prior CDK4/6 inhibitor.
* Undergone major surgery within 14 days of the initial dose of study drug
* Received another investigational agent (defined as any agent/device that has not received regulatory approval for any indication) within 14 days of the first dose of study drug for a nonmyelosupressive agent, or 21 days of the first dose of study drug for a myelosuppressive agent.
* Has any severe concurrent disease, infection, or comorbid condition that renders the patient inappropriate for enrollment in the opinion of the investigator.
* Has an active bacterial, fungal, and/or known viral infection. Patients with known HIV infection are excluded given the potential for interactions between antiretroviral agents and abemaciclib, and the potential for increased risk of life-threatening infection with therapy that is myelosuppressive. Patients with known Hepatitis B or Hepatitis C infection are excluded only if there is evidence of active infection (detectable Hepatitis B surface antigen, detectable Hepatitis C RNA)
* Documented brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with previously diagnosed brain metastases are eligible if they have completed treatment at least one month prior to trial registration, are neurologically stable, and have recovered from effects of radiotherapy or surgery.

  * Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks before the first study drug.
  * Treatment for brain metastases may have included whole brain radiotherapy, radiosurgery, or a combination as was deemed appropriate by the treating physician.
  * Patients who meet the above criteria and are clinically stable on anti-convulsant medication are eligible only if their anti-convulsant does not alter hepatic cytochrome P450 activity in a way that might interfere with metabolism of abemaciclib.
* Pregnant women are excluded from this study because of the potential for teratogenic effects.
* Lactating women are excluding from the study.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances: individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if they are diagnosed and have completed treatment within the past 5 years: cervical cancer in situ, and non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 5 years and felt to be at low risk of recurrence should be discussed with the principle investigator to determine eligibility.
* Have received any live vaccination within 28 days of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib: -Abemaciclib was administered orally, twice daily on days 1 to 28
  Abemaciclib: Abemaciclib (LY2835219) has been shown in vitro to be a selective ATP-competitive inhibitor of CDK4 and CDK6 kinase activity that prevents the phosphorylation and subsequent inactivation of the Rb tumor suppressor protein, thereby inducing G1 cell cycle arrest and inhibition of cell proliferation.
Period: Overall Study
Arm/Group | Abemaciclib
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abemaciclib
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 80]
Age, Customized [Count of Participants; unit: Participants]
  Age at enrollment: Less than 50 years old | 5
  Age at enrollment: Over 50 years old | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 24
  Race: Black | 2
  Race: Other | 1
Number of metastatic sites [Median (Full Range); unit: sites] | 7 [3 to 11]
Number of prior lines of systemic therapy for metastatic disease [Count of Participants; unit: Participants]
  0 | 2
  1 | 4
  2 | 14
  3 | 7
(Neo)adjuvant therapy [Count of Participants; unit: Participants]
  Yes | 22
  No | 5
Number of patients recurred within 12 months of their adjuvant systemic therapy [Count of Participants; unit: Participants] | 15
Prior chemotherapies in any setting [Number; unit: participants]
  Anthracycline | 18
  Taxane | 22
  Eribulin | 4
Prior immune therapy for early stage or metastatic disease [Count of Participants; unit: Participants] | 12
BRCA1 or BRCA2 Mutation [Count of Participants; unit: Participants]
  Present | 4
  Absent | 19
  Not reported | 4
Site of metastasis --Lung [Count of Participants; unit: Participants] | 12
Site of metastasis --Liver [Count of Participants; unit: Participants] | 8
Site of metastasis --Bone [Count of Participants; unit: Participants] | 15
Site of metastasis --Brain [Count of Participants; unit: Participants] | 6
Site of metastasis --Skin [Count of Participants; unit: Participants] | 10
Site of metastasis --Lymph node [Count of Participants; unit: Participants] | 23

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Overall Response Rate(ORR) = (CR + PR)/sample size.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 27
Participants | 0
Statistical Analysis 1: Comparison: Abemaciclib; Test type: Other; Objective Response Rate = 0.0, 95% CI 2-sided [0.000 to 0.247]

2. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression (per Response Evaluation Criteria in Solid Tumors 1.1) or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Baseline to the earlier of progression (per Response Evaluation Criteria in Solid Tumors 1.1), date of death due to any cause, or date of last disease evaluation. Participants will be followed up up to 16.5 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 27
months | 1.94 [1.84 to 11.47]

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Time Frame: Baseline to date of death due to any cause, or at date last known alive.Participants will be followed once every 6 months until death.Those removed from protocol therapy for unacceptable adverse event(s) will be followed until resolution or stabilization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 27
months | 8.44 [4.57 to 15.57]

4. Secondary Outcome: Disease Control Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD); Disease control rate is defined as CR + PR + SD ≥ 16weeks
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 27
Participants | 6
Statistical Analysis 1: Comparison: Abemaciclib; Test type: Other; Disease Control Rate = 0.222, 95% CI 2-sided [0.086 to 0.423]

5. Secondary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD); Clinical benefit rate is defined as CR+PR+SD ≥ 24weeks
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 27
Participants | 4
Statistical Analysis 1: Comparison: Abemaciclib; Test type: Other; Clinical Benefit Rate = 0.148, 95% CI 2-sided [0.042 to 0.337]

ADVERSE EVENTS:
Time Frame: 4.1 years
Description: Serious Adverse Events were defined as Grade 2/3 unexpected events with treatment attribution of possibly/probably/definitely, Grade 4 unexpected events with treatment attribution of possibly/probably/definitely and all Grade 5 events. All remaining AEs are classified as Other AEs (OAE) including Grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all Grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets.
Arm/Group | Abemaciclib
All-Cause Mortality (participants affected / at risk) | 24/27
Serious Adverse Events (participants affected / at risk) | 10/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib (N=27)
Abdominal pain (Gastrointestinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 3
Pericardial effusion (Cardiac disorders) | 2
Platelet count decreased (Investigations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chest pain-cardiac (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Pain (General disorders) | 1
Presyncope (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib (N=27)
Anemia (Blood and lymphatic system disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 7
Bloating (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 21
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 15
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 19
Gait disturbance (General disorders) | 2
Pain (General disorders) | 5
Creatinine increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 7
Lymph node pain (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT03130439/Prot_SAP_000.pdf